CLINICAL TRIAL: NCT02624349
Title: Immunogenicity and Safety of Human Papilloma Virus Vaccine in Solid Organ Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Upton Allen, Chief, division of infectious diseases, department of pediatrics, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000037024
Record Dates: First submitted 2013-10-07; First posted 2015-12-08 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Late Complication From Kidney Transplant; Complication of Transplanted Liver; Human Papillomavirus-Related Carcinoma
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transplant (Active Comparator): Intervention: Quadravalent human papillomavirus vaccine 0.5ml intramuscular injection at 0, 2, and 6 months and/or post administration antibody titers as described in methods
  Interventions: Drug: Quadravalent human papillomavirus vaccine
- Control (Active Comparator): Intervention: Quadravalent human papillomavirus vaccine 0.5ml intramuscular injection at 0, 2, and 6 months and/or post administration antibody titers as described in methods
  Interventions: Drug: Quadravalent human papillomavirus vaccine

INTERVENTIONS:
Drug: Quadravalent human papillomavirus vaccine — Vaccine will be administered to all transplant recipients. Controls will be recruited based on previous documented receipt of vaccine
  Other Names: Gardasil

SUMMARY:
The human papilloma virus (HPV) is known to be an important cause of cervical and anal cancers. Studies on patients who have received a solid organ transplant (such as a liver or kidney transplant) have suggested the risk of HPV-related cancers may be higher in this population. The HPV vaccine, Gardasil®, has been approved for use in males and females by Health Canada. In studies on healthy subjects this vaccine is nearly 100% effective at preventing infections from HPV serotypes that are in the vaccine. These serotypes, representing different viral strains, are known to cause 70% of cervical cancers and 90% of genital warts. The vaccine was also shown to be very safe and well tolerated in healthy subjects. Transplant patients are at higher risk of HPV related complications and cancers. As a result transplant experts have recommended this vaccine for use in their patients; however there have been no studies looking at the response to vaccination or safety of this vaccine in solid organ transplant recipients. Our objective is to study the immune response and side effects of Gardasil® in children who have received kidney or liver transplants. We will study this by comparing immune responses to the vaccine in healthy adolescent females compared to female liver and kidney transplant recipients. We will be recruiting females ages 12-19, as the province of Ontario funds the vaccine for this group. We will evaluate the transplant subjects for side effects after they receive the vaccine. Our hypothesis is that transplant recipients will have lower immunogenicity than healthy controls.

DETAILED DESCRIPTION:
1. Hypothesis The Human papillomavirus (HPV) vaccine, Gardasil®, will likely provide protection in solid organ transplant patients against the vaccinated strains with lower immunogenicity rates compared to healthy controls. We expect higher levels of immune suppression to influence immunogenic response.
2. Objective Primary: To evaluate the immunogenicity of the recombinant HPV vaccine, Gardasil®, in pediatric solid organ transplant recipients compared to controls, as well evaluate for clinical risk factors associated with lower responses in transplant recipients. Immunogenicity will be assessed through geometric mean titres (GMT) as well as seroconversion.

   Secondary: To evaluate the safety of Gardasil® in transplant recipients.
3. Background

   3.1 Disease HPV is known to predispose to cervical, anal, and a variety of head and neck cancers in both healthy adults and in those who are immunocompromised, including those who have received solid organ transplants. An estimated 3 million women in Canada are infected with HPV. Peak incidence occurs within 5-10 years of first sexual experience and adolescent females represent the largest cohort affected by HPV.

   3.2 Vaccine In 2006 the Food and Drug Administration approved the quadravalent recombinant HPV vaccine, Gardasil®, which targets strains 16 and 18 as well as 6 and 11, which are responsible for 70% of cervical cancer cases and 90% of genital warts, respectively. Health Canada has recently approved Gardasil® for use in females' aged 9-45 years and males 9-26 years. Gardasil® has been shown in numerous clinical trials to be effective in the management of HPV by preventing vaccine sub-type related infections and precancerous lesions. Gardasil® is regarded as generally safe and well tolerated based on reported adverse events through government databases in the United States, as well as analyses by independent researches. The bivalent HPV vaccine, Cervarix®, also appears safe and effective in preventing cervical cancer, however the data are less robust and there would be no protection against genital wart strains. Long term benefits of HPV vaccination are unknown, however models have predicted both a significant mortality benefit by preventing cases of cervical cancer7 and overall cost-effectiveness; particularly if the vaccine is administered to girls under the age of twelve.

   3.3 HPV in Transplant Patients Due to the prominent role of cell-mediated immunity in HPV, transplant recipients are felt to be at increased risk of infection leading to extensive or frequent warts, and increased incidence of skin and anogenital malignancies. Skin cancers are the most common malignancy affecting patients post transplantation. Anogenital cancer incidence is estimated to be 30-100 times greater in transplant patients compared to the general population. HPV is a preventable cause of a large number of these malignancies, suggesting that a vaccine could potentially thwart some of the morbidity and mortality experienced by transplant recipients. Furthermore, studies have suggested that organ transplant patients are more likely to be infected with HPV as well as develop secondary neoplasias. For these reasons vaccinating this population against HPV has the potential for significant long-term benefits.
4. Methods 4.1 Design We are proposing a prospective observational study by evaluating the serological response for the vaccine covered HPV serotypes; 6, 11, 16, and 18. This study will take advantage of routine, provincially funded population based vaccination program, and patients will receive the vaccine in the study that healthy adolescents receive at school in grades 7 or 8. Study subjects will be identified using the liver and kidney transplant clinical database and control subjects will be identified through the Hospital for Sick Children adolescent medicine clinic. A letter of introduction will be sent to the families. Consent will be obtained by the transplant nurse or physician known to the patient. Transplant subjects will undergo baseline and post-immunization serology to evaluate both GMT as well as to document seroconversion response to the vaccine. Gardasil® will be funded through the province of Ontario. Controls will receive their vaccine through the adolescent clinic, schools, or Toronto Public Health clinics in the community as per the recommended schedule. At recruitment attempt will be made to draw baseline serology status, vaccinate, and then collect post-immunization serology to document seroconversion. However, to facilitate recruitment for controls that have documented receipt of three doses of the vaccine these children will be recruited for post-vaccination serology only to compare GMTs. Control vaccines will also be funded by the province of Ontario and administered in accordance with Health Canada standards.

4.2 Investigational Agent

4.2.1 Vaccine storage and characteristics Gardasil® (Merck Canada Inc), the Quadravalent Human papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine, was selected for this study for its efficacy and safety data in healthy subjects, being publically funded by the province of Ontario, and it provides protection for 4 HPV serotypes. Gardasil® should be stored refrigerated 2-8 degrees Celsius, should not be frozen and remain protected from light. The total time outside of refrigerator should not to exceed 72 hours. Vaccines will be stored compliant with the division 5 Canadian regulations.

4.2.2 Administration of vaccine Gardasil® vaccine is recommended to be administered intramuscularly in deltoid or thigh at a dose of 0.5ml at 0, 2, and 6 months. While every effort will be made to keep the aforementioned schedule, studies support some flexibility in the schedule. The 2nd dose will be administered at least 1 month after the 1st, but not more than 9 months. The 3rd dose can be administered 3 months following the second dose, but not more than 1 year following the first dose. All 3 doses must be administered within a 1 year period to be included in analysis. Subjects will be monitored for 15 min post-vaccination for any adverse effects.

4.3 Sample Size The study will be powered based on GMT immunogenicity. Based on this primary outcome, we wish to compare serum titres in transplant patients compared with controls. The sample size calculation is based on 90% power and 95% confidence and the assumption that a HPV vaccination will result in protective titres in 80% of transplant patients compared to 100% of controls. A sample size of approximately 75 transplant recipients and 75 controls will therefore be preferred to detect a significant difference, however recruitment of at least 50 participants in each group is acceptable. Recruitment will take place over a 6 month period, resulting in a total study duration of approximately 12 months, up to a maximum of 18 months accounting for possible delays in vaccine administration up to 1 year from end of recruitment.

4.4. Analysis In the primary analysis of immunogenicity, the GMTs will be summarized for transplant recipients and compared with controls. The proportions of subjects achieving protective GMTs, as defined previously, will be compared using Chi-square or Fishers' exact test as appropriate. Means will be compared using Students t-test or a non-parametric procedure will be used to compare medians, as appropriate. Subjects and controls will be evaluated as a head-to-head comparison. For controls serology will be interpreted relative to time from last dose given. The investigators will use a multivariate analytic procedure to examine the effects of several independent variables with immunogenicity as the dependent variable. These independent variables are ones that could be potentially associated with differences in immune responsiveness (e.g., the interval between transplantation and vaccine administration). Other variables include the following: age; type of organ transplanted; presence or absence of graft rejection; type of immune suppression (e.g., use of anti-T lymphocyte therapy); immune globulin therapy; cytomegalovirus infection and disease; Epstein-Barr virus infection and disease; presence of bacterial opportunistic infections, concurrent diseases, steroid doses, and total lymphocyte count.

The secondary analysis will capture and describe the adverse effects among transplant recipients through telephone calls at 48 hours and 7 days utilizing the Public Health Ontario adverse event reporting form

4.5 Data Safety Monitoring Board and Research Ethics The study will be done with the approval of the institution's Research Ethics Board. In addition, although we have no reasons to anticipate problems with this vaccines in transplant patients, we will establish a Data Safety Monitoring Board that will review emerging data that relate to any major or catastrophic events that are temporally associated with the vaccine (even in the absence of obvious causality).

4.5.1 Early Termination or Withdrawal Subjects and/or parents/legal guardians have the right to withdraw from the study at any time for any reason. The investigator also has the right to withdraw subjects from the study if it is in the best interest of the subject.

Subject withdrawal criteria are as follows:

* Withdrawal of informed consent (subject's decision to withdraw for any reason)
* Serious adverse event which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject
* Any clinical adverse event or inter-current illness which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the subject (ex. Participants who develop symptoms of hypersensitivity after receiving the first or second dose of Gardasil® will be withdrawn from the study and will not receive further doses of Gardasil®)
* Pregnancy
* Subject non-adherence with the vaccine administration schedule defined above In the event a subject is withdrawn due to an Adverse Event, this will be recorded and subjects will continue to be followed until these events are resolved or stabilized, if possible.

4.5.2 Adverse Events All adverse events will be reported to the Hospital for Sick Children Research Ethics Board according to the Hospital for Sick Children's adverse event reporting requirements. All serious, unexpected adverse drug reactions to the study medication will be reported to Health Canada within 15 calendar days or for death or life-threatening events, within 7 calendar days. In the latter case, a follow-up report must be filed within 8 additional calendar days. Adverse reactions will be managed according to the Hospital for Sick Children's standard clinical management practices.

ELIGIBILITY:
Inclusion Criteria:

- Females 12-19 years of age

Exclusion Criteria

* Received transplant within the previous 6 months
* Males
* Pregnant
* Previous allergic reaction to any of the vaccine components
* Inadequate documentation of prior immunization

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity (Serum anti-HPV 6, 11, 16, and 18 antibody measured using a competitive Luminex immunoassay) | 4-6 weeks
  Serum anti-HPV 6, 11, 16, and 18 antibody will be measured using a competitive Luminex immunoassay (cLIA; reported in milli-Merck Units/ml). Seropositivity will be defined as an anti-HPV titre ≥20, 16, 20, and 24/ml, for HPV types 6, 11, 16, and 18, respectively

SECONDARY OUTCOMES:
Immunogenicity (Serum anti-HPV 6, 11, 16, and 18 antibody measured using a competitive Luminex immunoassay) | 1 year
  Serum anti-HPV 6, 11, 16, and 18 antibody will be measured using a competitive Luminex immunoassay (cLIA; reported in milli-Merck Units/ml). Seropositivity will be defined as an anti-HPV titre ≥20, 16, 20, and 24/ml, for HPV types 6, 11, 16, and 18, respectively

OTHER OUTCOMES:
Adverse event following immunization (AEFI) | 48 hours and 1 week
  phone calls will be made at 48hrs and 7 days to evaluate for any adverse events. The Public Health Ontario AEFI form will be used to identify local reactions, fevers, neurological complaints, and other temporally associated events. Any identified reactions are then quantified by severity and duration as indicated on the form. Adverse events will be qualitatively described.

CONTACTS AND LOCATIONS:
Overall Officials: Upton Allen, MD MSc, Principal Investigator — The Hospital for Sick Chidren
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No